CLINICAL TRIAL: NCT03466099
Title: A Randomized Sham-controlled Double-masked Phase 2a Study of the Efficacy, Safety and Tolerability of the Intravitreal Plasma Kallikrein Inhibitor, KVD001, in Subjects With Center-involving Diabetic Macular Edema Who Have Had Prior Anti-vascular Endothelial Growth Factor Treatment
Brief Title: Study of the Intravitreal Plasma Kallikrein Inhibitor, KVD001, in Subjects With Center-involving Diabetic Macular Edema (ciDME)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: KalVista Pharmaceuticals, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KVD001-201
Record Dates: First submitted 2018-02-26; First posted 2018-03-15 (Actual); Results first posted 2020-12-08 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Diabetic Macular Edema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- KVD001 Injection (high dose) (Experimental)
  Interventions: Drug: KVD001 Injection
- KVD001 Injection (low dose) (Experimental)
  Interventions: Drug: KVD001 Injection
- Sham Procedure (Sham Comparator)
  Interventions: Other: Sham Procedure

INTERVENTIONS:
Drug: KVD001 Injection — Intravitreal KVD001 Injection
  Other Names: KVD001
  Arms: KVD001 Injection (high dose); KVD001 Injection (low dose)
Other: Sham Procedure — Sham Procedure
  Arms: Sham Procedure

SUMMARY:
This is a clinical study where patients with diabetes and a vision threatening eye condition called "Diabetic Macular Edema" receive four injections into the eye at monthly intervals. The patients will already have tried the standard of care without complete success. The patients will be randomized to receive either a high dose, a low dose or a sham control treatment. The study will evaluate whether the new treatment improves vision and whether it changes the underlying course of the disease in the eye.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Type I or Type II diabetes mellitus (DM).
* BCVA of ≥19 letters (~20/400) and ≤73 letters (~20/40) in the study eye and ≥34 letters(~20/200 or better) in the fellow eye.
* Presence of ciDME in the study eye defined as CST ≥305 μm in women and ≥320 μm in men
* Subjects first anti-VEGF injection in the study eye occurred ≤36 months.
* Subjects have received at least 3 anti-vascular endothelial growth factor (VEGF) injections in the study eye within a 6-month period.
* The last anti-VEGF injection in the study eye is ≥ 8 weeks.

Exclusion Criteria:

* Evidence of ocular pathology (e.g. visually significant cataract) that impacts subject's vision in the study eye from any cause other than DME.
* Evidence/presence of amblyopia, vitreomacular traction, epiretinal membrane, foveal atrophy, or foveal ischemia, or any other condition in the macula that is thought to impair the subject's vision (other than DME).
* Prior treatment with panretinal photocoagulation or focal grid macular photocoagulation in the study eye within the previous 3 months.
* Prior treatment with intravitreal (IVT) steroid in the study eye (in the previous 3 months for triamcinolone, previous 6 months for Ozurdex and at any time for Iluvien).
* Prior treatment with topical NSAIDs or topical steroids in the study eye within 1 month.
* Prior treatment with systemic corticosteroids or systemic anti-VEGF therapy within 3 months.
* Prior vitrectomy in the study eye.
* Prior intraocular surgery in the study eye except for cataract surgery. Cataract surgery within the previous 6 months in the study eye is excluded.
* Intraocular pressure (IOP) of >22 mmHg in the study eye or use of >2 antiglaucoma agents (combination agents count as 2 agents) in the study eye.
* Evidence of infectious dacrocystitis, significant blepharitis, active conjunctivitis, infectious keratitis, or scleritis in either eye, or any other condition that might affect the safety of the IVT injection.
* Current active proliferative diabetic retinopathy (PDR), active anterior segment neovascularization (ASNV), active retinal neovascularization, or the presence of vitreous hemorrhage in the study eye.
* Poorly controlled DM.
* Uncontrolled hypertension
* Prior treatment with ocriplasminin the study eye within 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2018-02-16 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — KalVista Pharmaceuticals
Locations (31):
- United States (31):
  - KalVista Investigative Site, Phoenix, Arizona
  - KalVista Investigative Site, Tucson, Arizona
  - KalVista Investigative Site, Arcadia, California
  - KalVista Investigative Site, Beverly Hills, California
  - KalVista Investigative Site, Palm Desert, California
  - KalVista Investigative Site, Palo Alto, California
  - KalVista Investigative Site, Sacramento, California
  - KalVista Investigative Site, Santa Ana, California
  - KalVista Investigative Site, Tustin, California
  - KalVista Investigative Site, Golden, Colorado
  - KalVista Investigative Site, Fort Myers, Florida
  - KalVista Investigative Site, Miami, Florida
  - KalVista Investigative Site, Pensacola, Florida
  - KalVista Investigative Site, Winter Haven, Florida
  - KalVista Investigative Site, Augusta, Georgia
  - KalVista Investigative Site, Marietta, Georgia
  - KalVista Investigative Site, Indianapolis, Indiana
  - KalVista Investigative Site, Boston, Massachusetts
  - KalVista Investigative Site, Henderson, Nevada
  - KalVista Investigative Site, Lynbrook, New York
  - KalVista Investigative Site, Rochester, New York
  - KalVista Investigative Site, Cincinnati, Ohio
  - KalVista Investigative Site, Rapid City, South Dakota
  - KalVista Investigative Site, Abilene, Texas
  - KalVista Investigative Site, Arlington, Texas
  - KalVIsta Investigative Site, Austin, Texas
  - KalVista Investigative Site, Dallas, Texas
  - KalVista Investigative Site, Fort Worth, Texas
  - KalVista Investigative Site, San Antonio, Texas
  - KalVista Investigative Site, Charlottesville, Virginia
  - KalVista Investigative Site, Silverdale, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 130 Patients were randomized but one patient withdrew prior to receiving any study treatments
Groups:
- KVD001 Injection (High Dose): KVD001 Injection: Intravitreal KVD001 6μg Injection administered to the study eye on Day 1 and Weeks 4, 8 and 12.
- KVD001 Injection (Low Dose): KVD001 Injection: Intravitreal KVD001 3μg Injection administered to the study eye on Day 1 and Weeks 4, 8 and 12.
- Sham Procedure: Sham Procedure: Sham Procedure performed on the study eye on Day 1 and Weeks 4, 8 and 12 which involved preparing the study subject in the same manner as a real injection would be prepared (i.e., including but not limited to insertion of lid speculum, application of povidone-iodine, and subconjunctival injection of an anesthetic, all applied to the study eye) after which an empty syringe without an attached needle was pressed against the eye to mimic the pressure of an injection
Period: Overall Study
Arm/Group | KVD001 Injection (High Dose) | KVD001 Injection (Low Dose) | Sham Procedure
Started | 41 | 44 | 45 (One study subject consented and was randomized, but withdrew prior to receiving any study treatments)
Treated | 41 | 44 | 44
Completed | 24 | 30 | 28
Not Completed | 17 | 14 | 17
Not completed — Adverse Event | 1 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 3 | 1
Not completed — Use of rescue medication | 8 | 9 | 13
Not completed — Rescued without meeting criteria | 4 | 1 | 1
Not completed — Subject compliance | 2 | 0 | 0
Not completed — Worsening disease | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- KVD001 Injection (High Dose): KVD001 Injection: Intravitreal KVD001 Injection 6ug
- KVD001 Injection (Low Dose): KVD001 Injection: Intravitreal KVD001 Injection 3ug
- Total: Total of all reporting groups
Arm/Group | KVD001 Injection (High Dose) | KVD001 Injection (Low Dose) | Sham Procedure | Total
Number analyzed (Participants) | 41 | 44 | 44 | 129
Age, Categorical [Count of Participants; unit: Participants] — Age category by treatment group
  Participants
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 21 | 27 | 23 | 71
    >=65 years | 20 | 17 | 21 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (9.58) | 61.1 (10.67) | 64.6 (8.62) | 63.0 (9.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 20 | 23 | 58
  Male | 26 | 24 | 21 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 7 | 15 | 41
  Not Hispanic or Latino | 22 | 37 | 29 | 88
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 5 | 3 | 12
  White | 37 | 37 | 37 | 111
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Iris color [Count of Participants; unit: Participants]
  Black | 0 | 1 | 0 | 1
  Blue | 9 | 9 | 6 | 24
  Brown | 23 | 24 | 24 | 71
  Hazel | 7 | 7 | 11 | 25
  Green | 2 | 2 | 3 | 7
  Gray | 0 | 1 | 0 | 1
Baseline Height (cm) [Mean (Standard Deviation); unit: cm] | 167.98 (10.833) | 169.21 (11.579) | 164.78 (12.638) | 167.31 (11.788)
Baseline Weight (kg) [Mean (Standard Deviation); unit: kg] | 88.88 (13.605) | 94.94 (26.404) | 85.34 (20.139) | 89.74 (21.083)
Baseline BMI [Mean (Standard Deviation); unit: kg/(m*m)] | 31.71 (5.367) | 33.00 (7.728) | 31.58 (6.999) | 32.11 (6.778)

OUTCOME MEASURES:

1. Primary Outcome: BCVA
Description: Change from Baseline in Best Corrected Visual Acuity (BCVA)
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | KVD001 Injection (High Dose) | KVD001 Injection (Low Dose) | Sham Procedure
Number analyzed (Participants) | 40 | 44 | 44
Letters | 0.8 (6.65) | -0.3 (8.36) | -1.8 (12.27)

2. Secondary Outcome: DRSS
Description: Assessments of Diabetic Retinopathy Severity Score (DRSS, scale 10-85) to evaluate the percentage of eyes with a ≥2 step reduction in score from the baseline retinopathy severity as graded from fundus photography. Minimum and maximum values of the DRSS are 10 and 85, with the low end of the scale indicating absence of retinopathy which, as the score increases, so does the severity of the retinopathy such that a score of 85 is indicative of advanced proliferative diabetic retinopathy
Time Frame: 16 weeks
Population: FAS Population with observed data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | KVD001 Injection (High Dose) | KVD001 Injection (Low Dose) | Sham Procedure
Number analyzed (Participants) | 29 | 31 | 29
percentage of participants | 0 [0 to 0] | 3.2 [0.1 to 16.7] | 0 [0 to 0]

3. Secondary Outcome: CST
Description: Assessments of Central Subfold Thickness (CST) - analysis of covariance of change from baseline in the study eye at week 16
Time Frame: 16 weeks
Population: FAS Population with LOCF
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | KVD001 Injection (High Dose) | KVD001 Injection (Low Dose) | Sham Procedure
Number analyzed (Participants) | 40 | 44 | 44
μm | 10.9 (104.67) | 2.3 (108.83) | 8.2 (123.90)

ADVERSE EVENTS:
Time Frame: 28 Weeks
Arm/Group | KVD001 Injection (High Dose) | KVD001 Injection (Low Dose) | Sham Procedure
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/44 | 0/44
Serious Adverse Events (participants affected / at risk) | 3/41 | 3/44 | 2/44
Other Adverse Events (participants affected / at risk) | 22/41 | 26/44 | 23/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KVD001 Injection (High Dose) (N=41) | KVD001 Injection (Low Dose) (N=44) | Sham Procedure (N=44)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Localized infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KVD001 Injection (High Dose) (N=41) | KVD001 Injection (Low Dose) (N=44) | Sham Procedure (N=44)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 3 (3)
Diabetic retinal oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Macular oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Eye Pain (Eye disorders) | 2 (2) | 3 (3) | 0 (0)
Retinal aneurysm (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Retinopathy (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 2 (2) | 4 (4)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Eyelid injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Blood glucose fluctuations (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Medication residue present (Investigations) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 3 (4) | 4 (5) | 3 (3)
Monocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 4 (4) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 1 (1) | 1 (1)
Catatact (Eye disorders) | 0 (0) | 0 (0) | 2 (3)
Eye irritation (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Ocular discomfort (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Vitreous detachment (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Conjunctival follicles (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Detachment of macular retinal pigment (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Foreign body sensation in eyes (Eye disorders) | 0 (0) | 1 (2) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Posterior capsule opacification (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal neovascularisation (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal vessel avulsion (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Tooth disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 1 (4) | 0 (0)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 1 (2)
Non-cardiac chest pain (General disorders) | 1 (2) | 0 (0) | 0 (0)
Chronic hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Allergy to arthropod bite (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Cellulitis staphylococcal (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 2 (2) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood potassium increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Blood triglycerides increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Intraocular pressure increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Optic nerve cup/disc ratio increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Urine albumin/creatinine ratio increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Disarthria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Mental status change (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-04-09): https://cdn.clinicaltrials.gov/large-docs/99/NCT03466099/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-07): https://cdn.clinicaltrials.gov/large-docs/99/NCT03466099/SAP_001.pdf